CLINICAL TRIAL: NCT00274404
Title: Randomized Study Assessing the Antiviral Activity and Safety of Valacyclovir in Primary Infectious Mononucleosis
Brief Title: Controlled Trial of Valacyclovir in Infectious Mononucleosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Minnesota Medical Foundation (Other); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0311M53430
Record Dates: First submitted 2006-01-06; First posted 2006-01-10 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Infectious Mononucleosis
Keywords: infectious mononucleosis; Epstein-Barr virus; valacyclovir; quantitative PCR
MeSH Terms: conditions — Infectious Mononucleosis; Epstein-Barr Virus Infections | interventions — Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: valacyclovir

SUMMARY:
The hypothesis is that an antiviral drug (valacyclovir) will reduce the amount of Epstein-Barr virus (EBV) in the mouths of university students with infectious mononucleosis (mono) while being a safe drug. Because EBV is the cause of mono, it is expected that reduction of the amount of virus could result in faster recovery from the disease.

DETAILED DESCRIPTION:
University of Minnesota students 18 years of age or older who are referred by the Boynton student health service during the first 7 days of infectious mononucleosis are eligible to participate. All of the subjects who enroll will be allowed to complete the study, but only the information from those students who truly have mono due to a primary infection with EBV as determined by laboratory tests will be used for the results. The students will be assigned by chance(randomized)either to receive the antiviral drug valacyclovir at a dosage of a 1 gram tablet every 8 hours for 14 days or no antiviral drug. Nine research clinic visits over 180 days are scheduled for clinical exams, histories, and collection of mouth and blood samples. The amount of EBV in the mouth and blood will be measured by a molecular virology research test called real-time TaqMan polymerase chain reaction. The severity of illness will be evaluated using a scale that measures the degree of physical activity and intensity of symptoms. The safety of the drug will be monitored by periodically checking the blood cell counts, and assessing liver and kidney function among other parameters. Personnel who do the lab work and analyze the data will not know the subjects' study drug assignments so that the data can be collected and analyzed objectively. The study will remain open to enrollment until 20 subjects with laboratory-confirmed primary EBV have been enrolled and followed for at least 2 weeks. The study will end when all subjects complete all scheduled study visits.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of infectious mononucleosis with onset no more the 7 days before enrollment; willingness to sign informed consent
* Willingness to provide blood and oral washing samples at regular intervals
* Females must have a negative urine pregnancy test and agree to use effective contraception (barrier or hormonal) for the first 30 days of the study if assigned to valacyclovir
* Corticosteroids are permitted only if prescribed by the subject's primary physisican for treatment of this acute disease

Exclusion Criteria:

* Previous history of mono
* Pregnant or breast feeding
* End-stage renal or liver disease
* Immunosuppressed due to underlying medical disease and/or immunomodulating medications prior to enrollment
* Onset of present illness >7 days ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-02; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who have at least a 100-fold (2log10) drop in the amount of EBV in their oral washes during the 14-day treatment period

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of valacyclovir
Evaluate the quantity of EBV in the oral washings
Correlate severity of illness with the amount of virus in the oral and blood compartments
Evaluate the areas under the viral load - time curves

CONTACTS AND LOCATIONS:
Overall Officials: Henry H Balfour, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Clinical Virology Clinic, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Balfour HH, Jr., Hokanson KM, Schacherer RM, Fietzer CM, Schmeling DO, Brundage RC. A controlled trial of valacyclovir in infectious mononucleosis. Presented at the 45th Interscience Conference on Antimicrobial Agents and Chemotherapy, Washington, DC, December 18, 2005. Abstract V1392
- See also: University of Minnesota Clinical Virology Programs website — http://cvp.umn.edu